CLINICAL TRIAL: NCT03588897
Title: The Impact of Oral Nutritional Supplements on the Nutritional Status of the Elderly - Randomised Clinical Trial.
Brief Title: The Impact of Oral Nutritional Supplements on the Nutritional Status of Elderly Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radoslaw Pach, MD, Ph D (Other)
Responsible Party: Sponsor-Investigator, Radoslaw Pach, MD, Ph D, Assisstant Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nutrition in Elderly RCT
Record Dates: First submitted 2018-07-01; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Nutrition Disorders in Old Age; Nutritional Supplement Toxicity; Elderly Infection
Keywords: nutritional status; Nutridrink; elderly nutrition

STUDY DESIGN:
Intervention Model Description: Normal diet versus normal diet + nutritional support in elderly patients
Oversight: FDA-regulated Device: No

ARMS (2):
- Normal Diet (No Intervention): Elderly patients receiving normal diet
- Nutritional Support (Experimental): Elderly patients receiving normal diet with nutritional support (Nutridrink Multi Fibre 2x100 ml per day)
  Interventions: Dietary Supplement: Nutridrink Multi Fibre

INTERVENTIONS:
Dietary Supplement: Nutridrink Multi Fibre — Dietary supplementation of 300 kcal for 14 days
  Arms: Nutritional Support

SUMMARY:
The study compares nutritional status of two groups elderly patient aged 65 and more. One group of the patients received nutritional support (Nutridrink Multi Fibre) for 14 days. Nutritional status of the patients were compared 2 months after the start of the intervention.

DETAILED DESCRIPTION:
The aim of the study was to compare nutritional status of two groups of elderly patients (> 65 years old). Total of 120 patients were randomly assigned into two groups. One group received normal diet whereas the second group received 300 kcal nutritional support (Nutridrink Multi Fibre 2x100 ml) between meals for 14 days. Two months after start of the intervention following examinations were performed:

* functional status of the patient (Barthel's scale, MMSE scale)
* nutritional status based on: weight, height, BMI; Mini Nutritional Assessment, plasma concentration of prealbumin, albumin, transferrin, total lymphocyte count.

The clinical status of the patient was evaluated based on clinical data on different organ infections. In addition costs of supplementary nutrition were taken into consideration.

ELIGIBILITY:
Inclusion Criteria:

* age > 65 and general status which enables compliance with study requirements
* Barthel's scale (Barthel scale = Barthel ADL index - an ordinal scale used to measure performance in activities of daily living) points 21-100
* MMSE (Mini Mental State Examination) points 24-30
* no use of laxatives

Exclusion Criteria:

* lack of consent
* neoplasms
* previous enteral nutrition
* Barthel's scale 0-20
* MMSE points 0-23
* BMI > 25
* laxatives

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
BMI of the elderly patients | 2 months
  BMI two months after start of the intervention
Prealbumin plasma concentration | 2 months
  Prealbumin concentration two months after start of the intervention
Albumin plasma concentration | 2months
  Albumin concentration two months after start of the intervention
Transferrin plasma concentration | 2 months
  Transferrin concentration two months after start of the intervention
TLC | 2 months
  Total lymphocyte count two months after start of the intervention

SECONDARY OUTCOMES:
Organ infections | 2 months
  Infection in any organ based on clinical data
Complications | 2 months
  Any complications associated with nutritional support
Functional status of the patient - Barthel's scale | 2 months
  Scores in Barthel's scale two months after start of the intervention
Functional status of the patient - MMSE scale | 2 months
  Scores in MMSE scale two months after start of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Scislo, MD PhD, Principal Investigator — Department of Clinical Nursery, Jagiellonian University

IPD SHARING:
Plan to Share IPD: No